CLINICAL TRIAL: NCT05005286
Title: Comparison of Microbiota Composition and Antimicrobial Property From Breastmilk of Mothers With and Without Pregnancy Vaginal Infections
Brief Title: Evaluation of Breastmilk Microbiota as a Function for Immunity
Status: Completed | Type: Observational
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Min-Tze LIONG, Professor, Universiti Sains Malaysia
Other Study IDs: USM/JEPeM/20090500
Record Dates: First submitted 2021-08-08; First posted 2021-08-13 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Vaginal Infection; Breastmilk Collection
Keywords: Breastmilk; Vaginal Infection; Immunity properties
MeSH Terms: conditions — Vaginitis; Breast Milk Expression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Human breastmilk samples will be collected in this study. The procedure of collecting sample is hands must be washed before milk expression, and nipples are cleaned with sterile water and alcohol swab. 15mL of fresh breast milk will be collected into a tube and stored at -20℃ until further analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Lactating women with vaginal infection during pregnancy as confirmed by past medical records
  Interventions: Other: Past history of vaginal Infections
- Group B: Lactating women without any vaginal infection during pregnancy

INTERVENTIONS:
Other: Past history of vaginal Infections — With or without vaginal infection during pregnancy
  Groups: Group A

SUMMARY:
The aim of this study is to evaluate the difference of breast milk microbiota between mothers with and without vaginal infections during pregnancy.

DETAILED DESCRIPTION:
The maternal microbiota is one of the relevant factors in the development of the infant's immune system, whereby the colonization of microbes in human begins at birth, when the newborn baby is exposed to maternal vaginal, gastrointestinal microbiota and as well as the microbes from the external environment. The neonatal intestine is colonized by symbiotic bacteria can be divided into four main steps; (i) acquisition of maternal vaginal, colonic, and skin flora at birth; (ii) introduction of oral feedings (breastfeeding or formula feeding); (iii) weaning; and (iv) acquisition of complete adult colonization.

Breastfeeding is associated with the protection of the infants from either infections or infection-related conditions, such as gastroenteritis, upper and lower respiratory tract infection, acute otitis media, urinary tract infection, neonatal septicaemia and necrotizing enterocoltis. The protection is through the combination of action of the breast milk components, such as maternal immunoglobulins, immunocompetent cells, or variety of anti-microbial compounds. Besides that, breast milk also contains prebiotic substances which may selectively stimulate the growth of limited number of beneficial bacteria in the gut.

A total number of 100 lactating mothers are needed for this study. Subjects will be recruited from HUSM Kubang Kerian, USM Main Campus Penang, and Institut Perubatan & Pergigian Termaju USM Penang. The subjects will be explained on all related information in the consent form prior to signing. The procedure of collecting sample is hands must be washed before milk expression, and nipples are cleaned with sterile water and alcohol swab. 15mL of fresh breast milk will be collected into a tube and stored at -20℃ until further analyses.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women
* Willing to commit throughout the experiment

Exclusion Criteria:

* Long term medication due to certain illnesses for over 3 months during pregnancy
* Gestational diabetes during pregnancy
* History of diabetes, coronary heart disease, and hypertension in life
* BMI before pregnancy above 24.9
* Consuming probiotic product during pregnancy
* Consuming probiotic product during lactation period

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from HUSM Kubang Kerian, USM Main Campus Penang, USM Kelantan and Institut Perubatan & Pergigian Termaju USM.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Breastmilk microbiota profiles | 6 months
  Differences in breastmilk microbiota profiles via pyrosequencing from breastmilk of women with or without history of vaginal infection during pregnancy

SECONDARY OUTCOMES:
Immuno-modulatory properties of breastmilk | 6 months
  Differences in breastmilk concentrations of immunity parameters such as immunoglobulins and cytokines from breastmilk of women with or without history of vaginal infection during pregnancy
Antimicrobial properties of breastmilk microbiota | 6 months
  Differences in antimicrobial properties against vaginal pathogens using breastmilk of women with or without history of vaginal infection during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Min T Liong, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Main Campus USM, George Town, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No